CLINICAL TRIAL: NCT02613312
Title: Chemotherapy Followed by Surgery and Neoadjuvant Hemothoracic Intensity Modified Radiation Therapy (IMRT) for Patients With Malignant Pleural Mesothelioma
Status: Terminated | Type: Observational
Why Stopped: Practice change in what is considered standard of care
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dennis Wigle, Principal Investigator, Mayo Clinic
Other Study IDs: 15-007645; NCI-2024-02057 (Registry Identifier: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Mesothelioma; Solitary Fibrous Tumor of the Pleura
MeSH Terms: conditions — Mesothelioma; Solitary Fibrous Tumor, Pleural

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine the response rate and overall survival in patients that have been diagnosed with mesothelioma and will undergo chemotherapy, surgery and intensity modified radiation therapy (IMRT) as part of their standard of care.

DETAILED DESCRIPTION:
The investigators will consent patients that have been diagnosed with mesothelioma and will undergo chemotherapy followed by surgery and then IMRT as their standard of care. The investigators will collect data from past and future medical records as well as data regarding their health status for their lifetime by reviewing life status, treatment status and CT scans.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides informed consent
* Subject is >18 years of age
* Subject is deemed competent for making medical decisions
* Subject is scheduled to undergo chemotherapy followed by surgery and then IMRT
* Subject is a surgical candidate
* A negative pregnancy test is required in women of child-bearing potential, as standard of care.

Exclusion Criteria:

•Subject is <18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving treatment at the Mayo Clinic Rochester that have been diagnosed with mesothelioma and will undergo chemotherapy followed by surgery and then IMRT as their standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2016-03-18 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | 2 years
  OS is defined as the length of time from study enrollment to death by any cause. Survival status of patients will be monitored every 6 months

SECONDARY OUTCOMES:
Progression free survival (PFS) as evidenced by CT scan review | 2 years
  PFS is defined as the length of time from study enrollment to the time of disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Wigle, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials